CLINICAL TRIAL: NCT00255645
Title: A Long-Term, Post-Treatment, Safety Follow-Up, Multi-Center Study in Patients With Type 2 Diabetes Mellitus From the GALLANT, GALLEX or ARMOR Studies.
Brief Title: G-PLUS (GALLANT, GALLEX and ARMOR - Post Treatment Follow-up Study)
Status: Terminated | Type: Observational
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Other Study IDs: D6160C00056; EudraCT No 2005-001373-97
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a long-term safety follow-up study to assess the post-treatment safety, at 12 and 24 months, in patients with type 2 diabetes after participation in the phaseII/III studies GALLANT, GALLEX and ARMOR. In addition, selected patients, including those with pre-defined laboratory or clinical findings, will have a 12-week post-treatment follow-up visit, including laboratory evaluation and adverse event recording.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who either completed at least 6 months in a previous treatment study GALLANT, GALLEX or ARMOR or met a pre-defined laboratory or clinical finding during participation in any of the said studies.

Exclusion Criteria:

* Received open-label treatment with tesaglitazar (since this is a post-treatment study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500
Dates: Start 2005-09; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstrasZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (543):
- United States (165):
  - Research Site, Birmingham, Alabama
  - Research Site, Columbiana, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Searcy, Arizona
  - Research Site, Sierra Vista, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Carlisle, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Carmichael, California
  - Research Site, Chula Vista, California
  - Research Site, Elk Grove, California
  - Research Site, Encinitas, California
  - Research Site, Encino, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Northridge, California
  - Research Site, Orange, California
  - Research Site, Pasadena, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Spring Valley, California
  - Research Site, Tustin, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hills, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Cooper City, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Plantation, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Berwyn, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Chicago Heights, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Sterling, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Waterloo, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Bossier City, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Cadillac, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Excelsior Springs, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, Rolla, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Dover, New Hampshire
  - Research Site, Hamilton, New Jersey
  - Research Site, Pleasantville, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Flushing, New York
  - Research Site, Manlius, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Olean, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Cheswick, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Warminster, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Morristown, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Midland, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Roseland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Gig Harbor, Washington
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Menomonee Falls, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Morón, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Salta, Salta Province
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Cairns
  - Research Site, Geelong
  - Research Site, Melbourne
  - Research Site, Perth
  - Research Site, Sydney
  - Research Site, Tasmania
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Braine-l'Alleud
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Merksem
  - Research Site, Sint-Gillis-Waas
  - Research Site, Steenokkerzeel
- Brazil (6):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (35):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Coquitlam, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Truro, Nova Scotia
  - Research Site, Windzor, Nova Scotia
  - Research Site, Bolton, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Hastings, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Napanee, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smith Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (9):
  - Research Site, Brno
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Semily
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Estonia (5):
  - Research Site, Paide
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
  - Research Site, Viljandi
- Finland (19):
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Imatra
  - Research Site, Jakobstad
  - Research Site, Joensuu
  - Research Site, Kauniainen
  - Research Site, Kokkola
  - Research Site, Kouvola
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Salo
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vaasa
  - Research Site, Vantaa
- France (41):
  - Research Site, Ambriere Les Vallees
  - Research Site, Angers
  - Research Site, Béziers
  - Research Site, Briey
  - Research Site, Broglie
  - Research Site, Château-Gontier
  - Research Site, Cremeaux
  - Research Site, Fontaine Saint Martin
  - Research Site, Gan
  - Research Site, Hyères
  - Research Site, Jarny
  - Research Site, La Garde
  - Research Site, La Seyne-sur-Mer
  - Research Site, Lambersat
  - Research Site, Laval
  - Research Site, Le Brusc
  - Research Site, Le Lavandou
  - Research Site, Lille
  - Research Site, Lomme
  - Research Site, Marignane
  - Research Site, Mars Da Tour
  - Research Site, Mayenne
  - Research Site, Metz
  - Research Site, Mondelange
  - Research Site, Montbrison
  - Research Site, Montpellier
  - Research Site, Montrevault
  - Research Site, Moûtiers
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Roanne
  - Research Site, Roquevaire
  - Research Site, Saint-Chamond
  - Research Site, Saint-Cyr
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Six-Fours-les-Plages
  - Research Site, Tantonville
  - Research Site, Tiercé
  - Research Site, Toulon
  - Research Site, Toulouse
- Germany (20):
  - Research Site, Aschaffenburg
  - Research Site, Beckum
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Ehrenberg
  - Research Site, Essen
  - Research Site, Gelnhausen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Hermaringen
  - Research Site, Künzing
  - Research Site, Langen
  - Research Site, Mannheim
  - Research Site, Marl
  - Research Site, Nürberg
  - Research Site, Pirna
  - Research Site, Rotenburg/Fulda
- Greece (2):
  - Research Site, Athens
  - Research Site, Piraeus
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin, N.T.
- Hungary (8):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Gy?r
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Siófok
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, New Delhi
- Indonesia (2):
  - Research Site, Jakarta
  - Research Site, Malang
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Rishon LeZiyyon
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (19):
  - Research Site, Arenzano
  - Research Site, Chiavari (GE)
  - Research Site, Chieri
  - Research Site, Florence
  - Research Site, Gubbio (PG)
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monteccio Emilia
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Pescara
  - Research Site, Piacenza
  - Research Site, Pistoia
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Scandiano
  - Research Site, Udine
- Latvia (7):
  - Research Site, Daugavpils
  - Research Site, Jēkabpils
  - Research Site, Madona
  - Research Site, Riga
  - Research Site, Sigulda
  - Research Site, Talsi
  - Research Site, Valmiera
- Research Site, Vilnius, Lithuania
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kubang Kerian, Kota Bharu
- Mexico (6):
  - Research Site, Guadalajara, Jalisco
  - Research Site, México, D.F.
  - Research Site, Nuevo León, Monterrey
  - Research Site, Torreón
  - Research Site, Veracruz, Veracruz
  - Research Site, Zapopan , Jalisco
- Netherlands (10):
  - Research Site, Beek en Donk
  - Research Site, Bennebroek
  - Research Site, Deurne
  - Research Site, Huizen
  - Research Site, Losser
  - Research Site, Nijverdal
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, The Hague
- Norway (24):
  - Research Site, Aursmoen
  - Research Site, Ås
  - Research Site, Bergen
  - Research Site, Elverum
  - Research Site, Enebakk
  - Research Site, Fredrikstad
  - Research Site, Hamar
  - Research Site, Haugesund
  - Research Site, Horten
  - Research Site, Hønefoss
  - Research Site, Inderøy
  - Research Site, Kongsberg
  - Research Site, Larvik
  - Research Site, Lena
  - Research Site, Lierskogen
  - Research Site, Lysaker
  - Research Site, Oslo
  - Research Site, Rolvsøy
  - Research Site, Rud
  - Research Site, Soerumsand
  - Research Site, Stavanger
  - Research Site, Straume
  - Research Site, Trondheim
  - Research Site, Østerås
- Philippines (6):
  - Research Site, Cebu City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (19):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice - Ochojec
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, P³ock
  - Research Site, Poznan
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Toruñ
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zielona Góra
- Portugal (5):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Elvas
  - Research Site, Lisbon
  - Research Site, Portalegre
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Research Site, Belgrade, Serbia and Montenegro
- Research Site, Singapore, Singapore
- Slovakia (17):
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Ilava
  - Research Site, Košice
  - Research Site, Kysucké Nové Mesto
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Prešov
  - Research Site, Šahy
  - Research Site, Trenčín
  - Research Site, Trnava
  - Research Site, Veľký Meder
  - Research Site, Žilina
- South Africa (7):
  - Research Site, Cape Town
  - Research Site, Chatsworth
  - Research Site, Durban
  - Research Site, Gauteng
  - Research Site, Houghton Gauteng
  - Research Site, Johannesburg
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Begonte (Lugo)
  - Research Site, Guissona (Lleida)
  - Research Site, Madrid
  - Research Site, San Sebastián de los Reyes
  - Research Site, San Vicente de Raspeig (Alicante)
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Villar Del Arzobispo (Valencia)
- Sweden (14):
  - Research Site, Åmål
  - Research Site, Borås
  - Research Site, Dalby
  - Research Site, Gothenburg
  - Research Site, Höganäs
  - Research Site, Malmo
  - Research Site, Mölndal
  - Research Site, Partille
  - Research Site, Skene
  - Research Site, Skrivarp
  - Research Site, Stenungsund
  - Research Site, Uddevalla
  - Research Site, Uppsala
  - Research Site, Vänersborg
- Switzerland (5):
  - Research Site, Bern
  - Research Site, Ilanz
  - Research Site, Lausanne
  - Research Site, Monthey
  - Research Site, Zurich
- Taiwan (3):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Taipei
- Research Site, Bangkok, Thailand
- United Kingdom (31):
  - Research Site, Aberdeen
  - Research Site, Atherstone
  - Research Site, Ayr
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Berks
  - Research Site, Birmingham
  - Research Site, Bolton
  - Research Site, Bucks
  - Research Site, Cardiff
  - Research Site, Co Antrim N Ireland
  - Research Site, Co. Wexford, Ireland
  - Research Site, Coventry
  - Research Site, Dublin
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Kent
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Pembrokeshire
  - Research Site, Plymouth
  - Research Site, Radstock
  - Research Site, Reading
  - Research Site, Shrewsbury
  - Research Site, Surrey
  - Research Site, West Midlands
  - Research Site, Wiltshire
  - Research Site, Wrexham
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City